CLINICAL TRIAL: NCT00193869
Title: A Pilot Randomised Comparison of Dexamethasone 96 mg Versus 16 mg Per Day for Malignant Spinal Cord Compression Treated by Radiotherapy
Brief Title: SuperDEX Trial (Comparison of Two Doses of Dexamethasone for Malignant Spinal Cord Compression Treated by Radiotherapy).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Trans Tasman Radiation Oncology Group (Other)
Collaborators: Cancer Council New South Wales (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TROG 01.05
Record Dates: First submitted 2005-09-11; First posted 2005-09-19 (Estimated); Last update posted 2007-05-10 (Estimated); Status verified 2007-05

CONDITIONS: Spinal Cord Compression From Neoplasm Metastasis
Keywords: Radiotherapy; Dose fractionation
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Dexamethasone

SUMMARY:
The study aimed to pilot the viability of a full scale randomised comparison of 2 steroid doses in malignant spinal cord compression, to establish safety of high dose dexamethasone in this setting in Australia, to test web registration and randomisation and to compare different functional outcome measures.

DETAILED DESCRIPTION:
Malignant spinal cord compression (MSCC) is an uncommon condition with an estimated annual incidence of 2.5 per 100,000. It is a dreaded complication of malignancy because of the severe impact paralysis and sphincter disturbance has on quality and duration of survival.

Rat models have demonstrated the effectiveness of high doses of steroids. Only three randomised controlled trials (RCTs) have been published. The first compared radiotherapy to laminectomy plus radiotherapy in a series of 29 patients and failed to show any significant differences The widespread commonly used dose of Dexamethasone in Australia at that time was 16 mg/24 hr and the main concern for implementing higher doses was the toxicity profile reported in the few small randomised comparisons available at the time.In view of the conflict between standard Australian practice versus published (overseas) guidelines, a randomised comparison was proposed in Australia. This study was a pilot study initiated to determine the viability of a large trial, to pilot the use of web technology for trial conduct and to determine clinically useful outcome measures apart from simple ambulation rates.

Comparisons: Patients randomised to receive either 16mg/24hr or 96mg/24hr dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

* Malignant spinal cord compression with at least one of pain, weakness, sensory disturbance or sphincter disturbance
* Histology not required if prior biopsy proven malignancy
* Any stage
* Age >16 years
* ECOG 1-3 prior to cord compression event
* Minimum power 1 of 5 point scale Must not be paraplegic
* Minimum expected survival 2 months
* Relevant minimum lab values
* Patients capable of childbearing using adequate contraception
* Written informed consent

Exclusion Criteria:

* Prior radiotherapy to within vertebral±one level affected by cord compression
* Prior treatment for spinal cord compression at the current level
* Histology is lymphoma or myeloma
* Power less than 1 of 5
* More than 12 hours after initiation of dexamethasone>4mg/24hr
* Pre-existing co-morbid conditions - peptic ulceration or cardiac failure
* Allergy to study medications
* Multilevel cord compression or meningeal carcinomatosis
* Pregnant or lactating

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2001-09; Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Satisfactory recruitment | Failure to accrue 30 patients in 15 months will initiate early closure of this study.
Acceptable steroid toxicity rate at 28 days with reference to baseline. | 28 days

SECONDARY OUTCOMES:
Ambulation rates at 1 month | 1 month
Barthel Index | Final analysis when all patients have been followed for 1 month
Functional Independence (FIM) | Final analysis when all patients have been followed for 1 month
Functional Improvement Score (FIS)within 2 weeks with reference to baseline | 2 weeks
Pain | Final analysis when all patients have been followed for 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Peter Graham, FRANZCR, Study Chair — St George Hospital
Locations (1):
- St George Hospital, Kogarah, New South Wales, Australia

REFERENCES:
- [Result] Graham PH, Capp A, Delaney G, Goozee G, Hickey B, Turner S, Browne L, Milross C, Wirth A. A pilot randomised comparison of dexamethasone 96 mg vs 16 mg per day for malignant spinal-cord compression treated by radiotherapy: TROG 01.05 Superdex study. Clin Oncol (R Coll Radiol). 2006 Feb;18(1):70-6. doi: 10.1016/j.clon.2005.08.015. PMID 16477923
- See also: Click here for more information about this study on the TROG official website — http://www.trog.com.au